CLINICAL TRIAL: NCT04328480
Title: The ECLA PHRI COLCOVID Trial
Brief Title: The ECLA PHRI COLCOVID Trial. Effects of Colchicine on Moderate/High-risk Hospitalized COVID-19 Patients.
Acronym: COLCOVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estudios Clínicos Latino América (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLCOVID version 2.0
Record Dates: First submitted 2020-03-30; First posted 2020-03-31 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Simple pragmatic randomized open controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local standard of care plus colchicine (Active Comparator): Local standard of care plus colchicine (specific dosage schedule)
  Interventions: Drug: Colchicine; Other: Local standard of care
- Local standard of care (Other): Local standard of care for COVID-19 SARS moderate / high-risk patients
  Interventions: Other: Local standard of care

INTERVENTIONS:
Drug: Colchicine — The colchicine dosage schedule will vary according to the following scenarios:
  1. In patients not receiving Lopinavir/Ritonavir
     * Loading dose of 1.5 mg followed by 0.5 mg after two hours (day 1)
     * The next day 0.5 mg bid for 14 days or until discharge.
  2. In patients receiving Lopinavir/Ritonavir
     * Loading dose of 0.5 mg (day 1)
     * After 72 hours from the loading dose, 0.5 mg every 72 hours for 14 days or until discharge.
  3. Patients under treatment with Colchicine that are starting with Lopinavir/Ritonavir
     * Dose of 0.5 mg 72 hours after starting Lopinavir/Ritonavir.
     * Continue with 0.5 mg every 72 hours for 14 days or until discharge.
  Only the oral route will be used except in the case of patients associated with mechanical ventilation or with contraindications to the oral route, in whom it will be administered by nasogastric tube.
  Other Names: Colchicina
  Arms: Local standard of care plus colchicine
Other: Local standard of care — Local standard of care for COVID-19 SARS moderate /high-risk patients

SUMMARY:
The ECLA PHRI COLCOVID Trial is a simple, pragmatic randomized open controlled trial to test the effects of colchicine on moderate/high-risk hospitalized COVID-19 patients with the aim of reducing mortality and/or new requirement for mechanical ventilation.

DETAILED DESCRIPTION:
Various anti-viral treatments are being tested in clinical trials worldwide. The World Health Organization (WHO) launched a simple,pragmatic worldwide open-label trial to test Remdesivir, Lopinavir/Ritonavir, Interferon and Hydroxychloroquine or Chloroquine.The most important complication of COVID-19 severe cases is respiratory failure from severe acute respiratory syndrome (SARS), the leading cause of mortality. Accumulating evidence suggests that patients with severe COVID-19 might have a cytokine storm syndrome, a hyperinflammatory syndrome characterized by a fulminant and fatal hypercytokinemia and multiorgan failure.

The proposed pathophysiological mechanism of cytokine storm and inflammatory cascade activation is based on evidence collected primarily during the SARS-CoV and MERS-CoV epidemics (with a significant increase in IL1B, IL6, IL12, IFNγ, IP10, TNFα, IL15, and IL17 among others). The data collected during the pandemic with COVID-19 also shows a significant increase in inflammatory cytokines (GCSF, IP10, MCP1, MIP1A, and TNFα, among others) in sicker patients admitted to intensive care. In the absence of effective treatments for the management of patients with COVID-19 and respiratory failure, the immunomodulatory and anti-inflammatory effect of colchicine on cytokines involved in the hyper-inflammatory state is postulated. Several lines of research worldwide are testing powerful anti-inflammatory drugs for the pandemic, with different options including steroids, cytokine blockers, and other potent anti-inflammatory agents. Steroids are partially contraindicated in viral infections.

Colchicine is a powerful anti-inflammatory drug approved for the treatment or prevention of gout and Familial Mediterranean Fever at doses ranging between 0.3 mg and 2.4 mg/day. Its mechanism of action is through the inhibition of tubulin polymerization, as well as through potential effects on cellular adhesion molecules and inflammatory chemokines. It might also have direct anti-inflammatory effects by inhibiting key inflammatory signalling networks known as inflammasome and pro-inflammatory cytokines. Additionally, evidence suggests that colchicine exerts a direct anti-inflammatory effect by inhibiting the synthesis of tumor necrosis factor alpha and IL-6, monocyte migration, and the secretion of matrix metalloproteinase-9. Through the disruption of the cytoskeleton, colchicine is believed to suppress secretion of cytokines and chemokines as well as in vitro platelet aggregation. All these are potentially beneficial effects that might diminish or ameliorate the COVID-19 inflammatory storm associated with severe forms of the disease. Importantly, in one contemporary trial low-dose colchicine administered to patients who survived from acute coronary syndrome shows a statistically significantly reduction of cardiovascular complications.

We have therefore designed in a simple, pragmatic randomized controlled trial to test the effects of colchicine on severe hospitalized COVID-19 cases with the aim of reducing mortality.

Sample size calculation:

A minimum sample size of 1200 patients will provide 80% power to detect a relative risk reduction of approximately 30% in the treated group if the assumed composite rate (new requirement of intubation and / or death) in the control group is about 24%.

The ECLA PHRI COLCOVID Trial allows randomization to another trial, specifically patients included in the trial might be (or not) randomized to an antithrombotic strategy.

ELIGIBILITY:
Inclusion Criteria (case definition)

* Consented adults (age ≥18 years) and
* COVID-19 suspicious and
* Admitted to hospital or already in hospital and
* COVID-19 suggestive symptoms (fever or febrile equivalent, loss of smell and taste, fatigue, etc.) that may be present or absent at randomization time and
* SARS (severe acute respiratory syndrome)

  * shortness of breath (dyspnea) or
  * image of typical or atypical pneumonia or
  * oxygen desaturation (SpO2 ≤ 93)

Exclusion criteria

* Clear indication or contraindication for the use of colchicine
* Pregnant or breastfeeding female.
* Chronic renal disease with creatinine clearance <15 ml/min/m2
* Negative PCR test for SARS-COV2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1279 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Composite outcome: New requirement for mechanical ventilation or death | 28 days post randomization
  Number of participants who require new intubation for mechanical ventilation or die
Mortality | 28 days post randomization
  Number of participants who die

SECONDARY OUTCOMES:
New requirement for mechanical ventilation or death from respiratory failure | 28 days post randomization
  Number of participants who require new intubation for mechanical ventilation or die from respiratory failure
New requirement for mechanical ventilation or death from non-respiratory failure | 28 days post randomization
  Number of participants who require new intubation for mechanical ventilation or die from non-respiratory failure
Mortality due to respiratory failure | 28 days post randomization
  Number of participants who die from respiratory failure
Mortality due to non-respiratory failure | 28 days post randomization
  Number of participants who die from non-respiratory failure
In hospital - Composite outcome | During hospitalization or until death, whichever comes first, assessed up to 28 days
  Number of participants who require intubation for mechanical ventilation or die
In hospital - Mortality | During hospitalization or until death, whichever comes first, assessed up to 28 days
  Number of participants who die
Composite outcome (New requirement for mechanical ventilation or death) evaluated in Non-intubated population | 28 days post randomization
  Number of participants who were not intubated at randomization and require new intubation for mechanical ventilation or die
Mortality evaluated in Non-intubated population | 28 days post randomization
  Number of participants who were not intubated at randomization and die
Mean WHO descriptive score of COVID-19 during hospitalization | During hospitalization or until death, whichever comes first, assessed up to 28 days
  Mean WHO descriptive score of COVID-19 in the active treatment group compared to the placebo group
Highest WHO descriptive score of COVID-19 during hospitalization | During hospitalization or until death, whichever comes first, assessed up to 28 days
  Mean highest WHO descriptive score of COVID-19 in the active treatment group compared to the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Diaz, MD, Principal Investigator — ECLA- ICR
Locations (1):
- Sanatorio Parque, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slobodnick A, Shah B, Krasnokutsky S, Pillinger MH. Update on colchicine, 2017. Rheumatology (Oxford). 2018 Jan 1;57(suppl_1):i4-i11. doi: 10.1093/rheumatology/kex453. PMID 29272515
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Yusuf S, Collins R, Peto R. Why do we need some large, simple randomized trials? Stat Med. 1984 Oct-Dec;3(4):409-22. doi: 10.1002/sim.4780030421. No abstract available. PMID 6528136
- [Background] McDermott MM, Newman AB. Preserving Clinical Trial Integrity During the Coronavirus Pandemic. JAMA. 2020 Jun 2;323(21):2135-2136. doi: 10.1001/jama.2020.4689. No abstract available. PMID 32211830
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Derived] Diaz R, Orlandini A, Castellana N, Caccavo A, Corral P, Corral G, Chacon C, Lamelas P, Botto F, Diaz ML, Dominguez JM, Pascual A, Rovito C, Galatte A, Scarafia F, Sued O, Gutierrez O, Jolly SS, Miro JM, Eikelboom J, Loeb M, Maggioni AP, Bhatt DL, Yusuf S; ECLA PHRI COLCOVID Trial Investigators. Effect of Colchicine vs Usual Care Alone on Intubation and 28-Day Mortality in Patients Hospitalized With COVID-19: A Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2141328. doi: 10.1001/jamanetworkopen.2021.41328. PMID 34964849